CLINICAL TRIAL: NCT04120025
Title: Effectiveness of Diaphragmatic Breathing on Reflux Symptoms in Outpatients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, C. Joseph Yelvington P.T., D.P.T., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-011131
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: GERD
Keywords: Reflux; Heartburn
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Subject will continue standard of care for GERD symptoms
- Treatment Group (Experimental): Subjects will continue with usual care but will also receive diaphragm training (belly breathing) instructions using verbal, visual and tactile cues for proper contraction of the diaphragm as a home program
  Interventions: Behavioral: Diaphragm Training

INTERVENTIONS:
Behavioral: Diaphragm Training — training on isolated abdominal breathing with proper effort and hold time to promote strengthening
  Arms: Treatment Group

SUMMARY:
Researchers are trying to determine if abdominal breathing exercises can reduce symptoms associated with GERD (Gastroesophageal reflux disease).

DETAILED DESCRIPTION:
Much like the pelvic floor controls urinary incontinence the "abdominal roof" made of the diaphragm appears to have the ability to control reflux. Other studies have had positive results but from extensive training of outpatients. Our population comes from ambulatory outpatients from family medicine at MCJ. After consent they fill out a reflux disease questionnaire (RDQ) a valid instrument for measuring symptoms of reflux. Subjects are educated on the basic concept of the study and then instructed in isolated diaphragm contraction breathing. once they are proficient they are asked to continue this program 3 x 10 repetitions, 3 times per day supplemented by 10 more repetitions after each meal to reduce post prandial symptoms.

Follow up is done at 1, 3 and 6 months and includes reassessment via the RDQ and an assessment of estimated volume of exercise compliance.

ELIGIBILITY:
Inclusion Criteria:

* Adults with complaints of GERD, reflux, and/or heartburn symptoms

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Reflux Disease Questionnaire (RDQ) | Baseline, 1 month, 3 month, 6 month
  Change in self-reported reflux disease questionnaire using questions to assess subject symptoms. Subjects are asked to answer 12 questions based on their symptoms over the past seven days for frequency and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Yelvington, DPT, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Jacksonville, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials